CLINICAL TRIAL: NCT02193724
Title: Feasibility, Validation and Differentiation of Induced Pluripotent Stem Cells Produced From Patients With Heritable Retinoblastoma
Brief Title: Feasibility of Generating Pluripotent Stem Cells From Patients With Familial Retinoblastoma
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: RETCELL
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Retinoblastoma
Keywords: Heritable Retinoblastoma; Familial Retinoblastoma; Pluripotent Stem Cells
MeSH Terms: conditions — Retinoblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin samples or peripheral blood samples to be used to generate pluripotent stem cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinoblastoma: Participants identified with heritable retinoblastoma will undergo a skin biopsy or blood draw to collect cells for processing and analysis.
  Interventions: Other: Skin Biopsy; Other: Blood Draw

INTERVENTIONS:
Other: Skin Biopsy — A very small skin sample will be taken from the participant's arm. This will only be performed while the patient is under sedation for clinical purposes (e.g. exam under anesthesia, MRI, or other procedure requiring sedation).
  Other Names: Punch Biopsy
Other: Blood Draw — About 1 teaspoon of blood will be drawn from the participant's arm or from a central line catheter if present. Blood collection will be done at the same time the participant has blood drawn for routine clinical care.
  Other Names: Blood Sample

SUMMARY:
The goal of this study is to determine if human RB1-deficient induced pluripotent stem cells (iPSCs) can produce retina, and, furthermore, can give rise to retinoblastoma in culture. This unique opportunity to study the initiation of retinoblastoma in the developing retina will shed light on the cell of origin for retinoblastoma and allow the investigators to study the earliest molecular and cellular events in retinoblastoma tumorigenesis.

OBJECTIVES:

* To establish the feasibility of producing induced pluripotent stem cells (iPSCs) from retinoblastoma patients with germline RB1 mutations (RB1-deficient iPSCs).
* To validate human RB1-deficient iPSCs by confirming karyotype, pluripotency and RB1 mutation.
* To differentiate the RB1-deficient iPSCs into retina as a model of the initiation of retinoblastoma in the developing retina.

DETAILED DESCRIPTION:
This is an observational study where a small skin cell sample or peripheral blood sample will be used to produce iPSCs. After RB1-deficient iPSCs are produced, their karyotype and RB1 mutation will be confirmed and their pluripotency will be tested by studying the expression of pluripotent genes and proteins according to standardized guidelines established for human iPSCs. After validation of the RB1-deficient iPSCs, they will be differentiated in the laboratory into retina following established protocols.

ELIGIBILITY:
Inclusion Criteria:

* Research participant with heritable retinoblastoma and one of the following criteria:

  * Family history with RB1 mutation identified
  * Diagnosis of bilateral retinoblastoma
  * Diagnosis of unilateral retinoblastoma with RB1 mutation or MYCN amplification identified
* Participant or legal guardian/representative is able and willing to provide written informed consent.

Exclusion Criteria:

* Participants who do not meet the inclusion criteria will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have a diagnosis of heritable retinoblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Number of samples which successfully produced iPSCs | Once at enrollment
  Skin biopsy or peripheral blood mononuclear cells will be collected from eligible, consenting participants and shipped directly to the University of Wisconsin for processing. All samples will be returned to the St. Jude investigator within two months of reprogramming for further analysis.

SECONDARY OUTCOMES:
Number of samples with validated RB1-deficient iPSCs | Once at enrollment
  Samples will be analyzed for standard G band karyotype and FISH analysis (RB1 probe), targeted RB1 mutation (based on known mutation of patient from whom the sample was derived), and validation of pluripotency based on standard protocols.
Number of samples that differentiate human iPSCs toward an eye field fate | Once at enrollment
  The best available methodology will be utilized for analyses of the RB1-deficient iPSCs.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C. Brennan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols